CLINICAL TRIAL: NCT07250477
Title: Risk-adapted, Proteomic-guided Systemic Therapy for Previously Untreated Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC323; NCI-2026-00133 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer Stage IIIC; Non-small Cell Lung Cancer Stage IV; Non Small Cell Lung Cancer; Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer Unresectable
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systemic immune checkpoint inhibitor (ICI)-based therapy informed by PROphet CB and CARG-TT (Experimental)
  Interventions: Drug: Systemic (ICI)-based therapy informed by the PROphet CB assay and the CARG-TT assessment.
- Standard of Care (Active Comparator): Standard of care (SOC) biomarker assessment and subsequent selection of SOC systemic therapy.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Systemic (ICI)-based therapy informed by the PROphet CB assay and the CARG-TT assessment. — Pretreatment assessment with PROphet CB and CARG-TT, which will be used to determine which first-line systemic treatment participants in the intervention arm receive. Systemic treatment will be pre-determined by the trial, according to the results from PROphet CB and CARG-TT.
  Arms: Systemic immune checkpoint inhibitor (ICI)-based therapy informed by PROphet CB and CARG-TT
Drug: Standard of Care — Standard of care (SOC) biomarker testing followed by first-line treatment with either anti-PD(L)1 Immune checkpoint inhibitor (ICI) monotherapy or anti-PD(L)1 ICI + chemotherapy.
  Arms: Standard of Care

SUMMARY:
This is a phase 2, pragmatic, 1:1 randomized, open-label study that evaluates risk-adapted, proteomic-guided systemic therapy to improve 12-month progression free survival (PFS) among patients with previously untreated advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
Participants will be randomized to an intervention arm or a standard of care (SOC) arm. Participants in the intervention arm will undergo pretreatment assessment with PROphet Clinical Benefit (CB) and the Cancer and Aging Research Group Toxicity Tool (CARG-TT); data from the assessments will be used to select systemic therapy, which can be any SOC treatment that incorporates a Programmed death-ligand 1 (PD-(L)1) antibody with or without chemotherapy and/or with or without Cytotoxic T-lymphocyte associated protein 4 (CTLA4) antibody. Participants in the SOC arm will undergo SOC biomarker assessment and subsequent selection of SOC systemic therapy. The primary endpoint is 12-month progression free survival (PFS). The findings will be stratified according to participant performance status and tumor PD-L1 score. The hypothesis is that risk-adapted, proteomic-guided systemic therapy will improve PFS among patients with previously untreated advanced NSCLC compared to SOC systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed non-small cell lung cancer that is metastatic or unresectable (stage IIIC or IV), deemed appropriate to receive standard of care immune checkpoint inhibitor-based therapy given with palliative intent.
* Age ≥18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥50%).
* Ability to understand and willingness to sign the informed consent form (ICF).
* Stated ability and willingness to adhere to all protocol requirements while on study

Exclusion Criteria:

* Tumor with known sensitizing alteration in ALK, EGFR, HER2, MET exon 14, NTRK, RET, or ROS1.
* Medical comorbidities precluding immune checkpoint inhibitor-based therapy per treating investgator's discretion.
* Previous systemic therapy for metastatic Stage IIIC or IV NSCLC. Patients who previously completed systemic therapy for early stage or locally advanced NSCLC ≥ 80 days prior to trial registration are eligible for inclusion.
* Any condition that in the opinion of the investigator would interfere with the participant's safety or compliance while on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2036-05 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate 12-month progression free survival (PFS) of systemic therapy informed by PROphet CB and CARG-TT (intervention arm) versus standard of care systemic therapy | Up to 12 months.
  Progression free survival (PFS) at 12 months, defined as progression assessed per investigator using Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 or death due to any cause at 12 months (± 28 days) from start of treatment.

SECONDARY OUTCOMES:
To evaluate treatment-related adverse events of systemic therapy informed by PROphet CB and CARG-TT (intervention arm) versus standard of care systemic therapy. | 3, 6, 9, and 12 months
  * Grade ≥3 treatment-related adverse events from chemotherapy classified and graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
  * Grade ≥2 treatment-related adverse events from immune checkpoint inhibitors classified and graded per NCI CTCAE v5.0
  * Number of dose delays, dose reductions, and/or dose discontinuations for treatment-related adverse event
  * Initiation and dose of systemic steroids for possible immune-related adverse event
To evaluate time to treatment discontinuation of systemic therapy informed by PROphet CB and CARG-TT (intervention arm) versus standard of care systemic therapy | Up to 12 months
  Time from the start of treatment to the date of treatment discontinuation or death due to any cause, whichever occurs first
To evaluate overall PFS of systemic therapy informed by PROphet CB and CARG-TT (intervention arm) versus standard of care systemic therapy. | Up to 60 months.
  Overall progression free survival (PFS) defined as the time from the start of treatment to the first date of the progression (any progression assessed per investigator using RECIST v1.1) or death due to any cause, whichever occurs first.
To evaluate overall survival (OS) among participants treated with systemic therapy informed by PROphet CB and CARG-TT (intervention arm) versus standard of care systemic therapy. | Up to 60 months.
  Overall survival (OS) defined as the time from the start of treatment to death due to any cause or 60 months, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Surbhi Singhal, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States